CLINICAL TRIAL: NCT03711383
Title: The Effects of Inulin on Acetate Production and Human Substrate Metabolism
Brief Title: Inulin and Acetate Production and Human Substrate Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL63754.068.17
Record Dates: First submitted 2018-07-06; First posted 2018-10-18 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Pre Diabetes
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Inulin; Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): isocaloric maltodextrin the day before CIDs
  Interventions: Dietary Supplement: Placebo
- Inulin (Active Comparator): 12 g of inulin + isocaloric maltodextrin the day before CID
  Interventions: Dietary Supplement: Inulin
- Inulin and Resistant Starch (Experimental): 12 g inulin + 7.5 g resistant starch the day before CID
  Interventions: Dietary Supplement: Inulin and Resistant Starch

INTERVENTIONS:
Dietary Supplement: Inulin and Resistant Starch — 12g per inulin in combination 7.5 g resistant starch per day the day before the CID Resistant starch 7.5 g
  Arms: Inulin and Resistant Starch
Dietary Supplement: Inulin — 12g per inulin in combination with maltodextrin per day the day before the CID
  Arms: Inulin
Dietary Supplement: Placebo — isocaloric maltodextrin before test day
  Arms: Placebo

SUMMARY:
Based on our hypothesis that orally administered resistant starch and inulin/beta glucan will be fermented into a SCFA pattern high in acetate and that this will lead to beneficial effects on human substrate and energy metabolism, we aim to address the following primary objective:

To investigate the effects of an acute administration of inulin/beta glucan in combination with resistant starch on fecal and plasma acetate, as well as on fasting and postprandial substrate and energy metabolism in lean normoglycemic men and obese, prediabetic men.

ELIGIBILITY:
Inclusion Criteria:

* lean (BMI ≥ 20kg/m2 and ≤ 24.9kg/m2)
* normoglycemic
* aged 30 - 65 years

OR

* overweight/obese (BMI ≥ 25kg/m2 and ≤ 34.9kg/m2)
* pre-diabetes
* aged between 30 - 65 years.

Exclusion Criteria:

* diabetes mellitus
* gastroenterological diseases or major abdominal surgery (allowed i.e.: - appendectomy, cholecystectomy)
* lactose intolerance and other digestive disorders
* cardiovascular disease, cancer, liver or kidney malfunction (determined -based on ALAT and creatinine levels, respectively)
* disease with a life expectancy shorter than 5 years
* Use of antibiotics 3 months prior inclusion
* Use of probiotics or prebiotics

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Plasma acetate concentrations (microM) | At baseline and up to four hours after a high-fat mixed meal of each CID

SECONDARY OUTCOMES:
Energy expenditure (in kJ/min) using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands) | At baseline and up to four hours after a high-fat mixed meal of each CID
Fat oxidation (in g/min) using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands) | At baseline and up to four hours after a high-fat mixed meal of each CID
Carbohydrate oxidation (in g/min) using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands) | At baseline and up to four hours after a high-fat mixed meal of each CID
Circulating hormone concentrations (Insulin, GLP-1, PYY) | At baseline and up to four hours after a high-fat mixed meal of each CID
Circulating metabolite concentrations (Glucose, Free Fatty Acids, Triglycerides) | At baseline and up to four hours after a high-fat mixed meal of each CID
Breath H2 using (Bedfont EC60 Gastrolyzer, Rochester, UK) | At baseline and up to four hours after a high-fat mixed meal of each CID

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Canfora EE, Hermes GDA, Muller M, Bastings J, Vaughan EE, van Den Berg MA, Holst JJ, Venema K, Zoetendal EG, Blaak EE. Fiber mixture-specific effect on distal colonic fermentation and metabolic health in lean but not in prediabetic men. Gut Microbes. 2022 Jan-Dec;14(1):2009297. doi: 10.1080/19490976.2021.2009297. PMID 34923911